CLINICAL TRIAL: NCT06476093
Title: SRT Combined With Anlotinib for the Treatment of Brain Metastases From Non-small Cell Lung Cancer: a Single-arm, Prospective, Exploratory Clinical Study
Brief Title: SRT Combined With Anlotinib for the Treatment of Brain Metastases From Non-small Cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Lianyungang (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-20231219001-01
Record Dates: First submitted 2024-06-10; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Non-Small-Cell Lung Cancer; Brain Metastases
Keywords: Anlotinib; SRT; Non-Small-Cell Lung Cancer; Brain Metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib+SRT Group (Experimental): Anlotinib#12mg#PO#Q3W#d1-14#
  Interventions: Drug: Anlotinib hydrochloride

INTERVENTIONS:
Drug: Anlotinib hydrochloride — Anlotinib#12mg#PO#Q3W#d1-14# SRT#depends
  Other Names: SRT

SUMMARY:
To evaluate the efficacy and safety of SRT combined with anlotinib in the treatment of limited brain metastases from non-small cell lung cancer.

DETAILED DESCRIPTION:
Anlotinib indication: Anlotinib is a novel oral multi-target receptor tyrosine kinase inhibitor, which has been shown to inhibit tumor growth by suppressing signaling pathways involving angiogenesis and cell proliferation. It has been approved by the Chinese National Medical Products Administration as a third-line therapy for NSCLC.

SRT indication: SRT（Stereotactic Radiation Therapy） is a form of local radiation therapy that delivers high doses of radiation in a limited number of treatments. Within Chinese guidelines and consensus, it is clearly defined that limited intracranial metastases can be treated with SRT instead of WBRT (Whole Brain Radiotherapy), achieving comparable or even superior efficacy while better preserving neurocognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in this study, sign informed consent, and demonstrate good compliance.
2. Patients with histologically or pathologically confirmed EGFR wild-type and EGFR mutant non-small cell lung cancer resistant to treatment.
3. The number of brain metastases is ≤ 5, and the patient has at least one assessable brain metastasis on imaging (RECIST 1.1). Additionally, the patient's physical condition allows for the completion of stereotactic radiosurgery.
4. Age between 18-80 years, gender unspecified.
5. ECOG performance status of 0 or 1; expected survival of no less than 3 months.
6. Regardless of prior treatment, it is only required that concurrent oral administration of anlotinib during radiotherapy without intervention regarding subsequent treatment regimens.
7. Oral administration of anlotinib including, but not limited to, third-line therapy.
8. Good function of major organs, with laboratory test indicators meeting the following criteria:

<!-- -->

1. Hematological examination:

   1. Hemoglobin (Hb) ≥ 90g/L (no blood transfusion within 14 days);
   2. Absolute neutrophil count (ANC) ≥ 1.5×10^9/L; total white blood cell count ≥ 3.5×10^9/L;
   3. Platelets (PLT) ≥ 100×10^9/L;
2. Blood biochemistry examination:

   a、Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (≤ 5 × ULN for liver metastasis/bone metastasis; ≤ 5 ULN for tumor bone metastasis); b、Total bilirubin (TBIL) ≤ 1.5 × ULN; c、Serum creatinine (Cr) ≤ 1.5×ULN or creatinine clearance rate ≥ 60 ml/min;
3. Coagulation function examination: Activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5×ULN.

   Exclusion Criteria:
   1. Squamous cell carcinoma patients (including adenosquamous carcinoma patients) should be excluded under the following conditions:

      ① Cavitary lung cancer.

      ② Patients who have had hemoptysis within the last month before the first dose and with a maximum daily hemoptysis of ≥2.5 mL, as well as other significant clinically relevant bleeding symptoms or those with a clear bleeding tendency combined with diseases/history.
   2. Patients with diffuse pleural metastases, malignant pericardial effusion, or diffuse spinal cord involvement.
   3. Patients with a history of other malignancies within 5 years (excluding cured basal cell carcinoma of the skin, prostate intraepithelial neoplasia, and cervical intraepithelial neoplasia).
   4. Current presence of pulmonary pneumonia with CTCAE 5.0 grade ≥ 2.
   5. Individuals with various factors that affect oral medication (such as dysphagia, gastrointestinal resection, chronic diarrhea, and intestinal obstruction).
   6. Evidence of active bleeding, or unexplained persistent decrease in hemoglobin. Screening/enrollment should be postponed until bleeding stops and the investigator deems it safe.
   7. Within the first 4 weeks before the initial dose, occurrence of any bleeding or hemorrhagic event ≥ Grade 3 according to CTCAE 5.0 standards; use of anticoagulants or vitamin K antagonists such as warfarin, heparin, or similar agents for treatment; under the condition that prothrombin time international normalized ratio (INR) ≤ 1.5, allowing the use of low-dose warfarin for prophylactic purposes (≤ 1mg/d), low-dose heparin (≤ 12,000 U/d), or low-dose aspirin (≤ 100mg/d).
   8. Within the 4 weeks before the initial dose, the presence of unhealed wounds, fractures, active ulcers of the stomach and duodenum, ulcerative colitis, or active bleeding from unresected tumors, or conditions judged by the investigator to potentially cause gastrointestinal bleeding or perforation; or patients who have undergone major surgeries (excluding vascular access surgery).
   9. Receipt of traditional Chinese medicine listed in the NMPA-approved drug instructions, which explicitly have indications for anti-tumor and lung cancer treatment (including compound Bupleurum capsules, Kangai injection, Conlear capsules/injections, Edaravone injections, Yadanzi oil injections/capsules, Xiaocanping tablets/injections, HuaChanSu capsules), or immune modulating drugs (excluding local use for pleural effusion control) within 2 weeks before the initial dose.
   10. History of organ or hematologic system transplantation.
   11. Presence of clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction.
   12. Patients with severe and/or uncontrolled diseases, including:

       * Patients with poorly controlled blood pressure (systolic blood pressure ≥150 mmHg, diastolic blood pressure ≥90mmHg);

         * Occurrence of thrombotic events, ischemic stroke, myocardial infarction within 6 months of the first dose, congestive heart failure of Grade ≥2, or requiring treatment for arrhythmias (including QTc ≥480ms);

           * Active or uncontrolled severe infections (grade ≥ 2 infection according to CTCAE 5.0), tuberculosis patients; ④ Known clinically significant liver disease history, including viral hepatitis, active HBV infection must be excluded for carriers of known hepatitis B virus (HBV) through positive HBV DNA (>2500 copies/mL or >500 IU/mL); known HCV infection and positive HCV RNA (>1×10^3 copies/mL), or other decompensated liver disease, chronic hepatitis requiring antiviral therapy; ⑤ Positive HIV test, positive rapid plasma reagin (RPR) test for syphilis; ⑥ Poorly controlled diabetes (fasting blood glucose ≥10mmol/L); ⑦ Urinalysis showing urinary protein ≥++, with confirmed 24-hour urinary protein quantification >1.0 g;
   13. According to the judgment of the principal investigator, patients with other factors that may lead to the forced termination of this study, such as other serious illnesses (including mental illness) requiring combined treatment, significant laboratory abnormalities, family or social factors affecting patient safety, or data and sample collection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
intracerebral Progression-Free-Surviva（iPFS） | 20 months
  The time from the start of treatment to intracranial tumor progression or death for any reason
  The time from the start of treatment to intracranial tumor progression or death for any reason
  The time from the start of treatment to intracranial tumor progression or death for any reason
intracerebral Objective Response Rate (iORR) | 20 months
  The proportion of patients whose intracranial tumor volume has reduced to a predetermined value and can maintain the minimum time limit

SECONDARY OUTCOMES:
intracerebral Progression-Free-Survival rate at 6 months and 1 year | 12 months
Progression-Free-Survival（PFS） | 20 months
Objective Response Rate（ORR） | 20 months
intracerebral Disease Control Rate（iDCR） | 20 months
Disease Control Rate（DCR） | 20 months
Overall Survival（OS） | 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Jiang, Doc, Study Chair — THE FIRST PEOPLE'S HOSPITAL OF LAINYUNGANG
Locations (1):
- The First People's Hospital of Lianyungang, Lianyungang, Jiangsu, China